CLINICAL TRIAL: NCT00738712
Title: Refinement and Assessment of New Magnetic Resonance Imaging (MRI) Technologies for Vascular, Abdominal, and Pelvic Exams
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: General Electric (Industry); Philips Healthcare (Industry)
Responsible Party: Principal Investigator, William Masch, Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00041815
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: Vascular MRI; Abdominal MRI; Pelvic MRI; Breast MRI; Magnetic Resonance Imaging (MRI)
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- New MRI techniques (Experimental): New hardware or software technologies designed to improve MRI (Magnetic Resonance Imaging) exams.
  Interventions: Procedure: MRI Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: MRI Magnetic Resonance Imaging — MRI
  Other Names: Magnetic Resonance Imaging

SUMMARY:
This study is being done to assess new Magnetic Resonance Imaging (MRI) technologies designed to improve MRI examinations of the vascular structures, abdomen, and pelvis regions.

DETAILED DESCRIPTION:
This study is being done to assess new Magnetic Resonance Imaging (MRI) technologies such as new hardware or software designed to improve MRI examinations of the vascular structures, abdomen, and pelvis regions. Software and hardware are always being improved, new machines replace old machines, software is updated and improved as well as devices used to produce better MRI images.

ELIGIBILITY:
Inclusion Criteria:

* male or non-pregnant female patient
* 18 years or older
* any ethnic background
* presenting to MRI for a clinically-ordered chest MRI exam.

Exclusion Criteria:

* Patients, who have electrically, magnetically or mechanically activated implants such as heart pacemaker, magnetic surgical clips, prostheses or implanted neurological stimulator.
* Pregnant patients or patients who are lactating.
* A patient who is claustrophobic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-05-02 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Evaluation of new software in MRI vascular imaging | 1 year
  New software technology will be utilized to enhance MRI imaging of the vascular regions of the body.

CONTACTS AND LOCATIONS:
Overall Officials: William Masch, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No